CLINICAL TRIAL: NCT03277599
Title: Ultrasound Guided Superficial Cervical Plexus Block Versus Greater Auricular Nerve Block for Tympanomastoid Surgery Pain
Brief Title: Comparison of Two Pain-treatment Techniques After Tympanomastoid Surgery Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2016/21-02
Record Dates: First submitted 2017-07-17; First posted 2017-09-11 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Pain Management; Nerve Block; Ultrasound
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Tramadol

STUDY DESIGN:
Intervention Model Description: prospective,randomized,single blind
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup Y (Active Comparator): ultrasound guided superficial cervical plexus blockage with 10 ml % 0.25 bupivacaine+IV patient-controlled analgesia (PCA) tramadol
  Interventions: Drug: IV patient-controlled analgesia (PCA) tramadol; Drug: ultrasound guided superficial cervical plexus block
- Grup B (Active Comparator): ultrasound ultrasound guided Great Auricular nerve blockage with 5 ml % 0.25 bupivacaine +IV patient-controlled analgesia (PCA) tramadol
  Interventions: Drug: IV patient-controlled analgesia (PCA) tramadol; Drug: ultrasound guided Great Auricular nerve block

INTERVENTIONS:
Drug: IV patient-controlled analgesia (PCA) tramadol — Tramadol infusion (PCA): 400 mg tramadol, IV 4 mg/mL tramadol solution into 100 mL normal saline; PCA settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Other Names: Tramadol
Drug: ultrasound guided superficial cervical plexus block — ultrasound guided superficial cervical plexus blockage with 10 ml % 0.25 bupivacaine
  Other Names: superficial cervical plexus block
  Arms: Grup Y
Drug: ultrasound guided Great Auricular nerve block — ultrasound guided Great Auricular nerve blockage with 5 ml % 0.25 bupivacaine +IV patient-controlled analgesia (PCA) tramadol
  Other Names: Great Auricular nerve block
  Arms: Grup B

SUMMARY:
Analgesia following tympanomastoid surgery is critical for the prevention of postoperative . There are very few regional anesthesia methods used to achieve this goal.

DETAILED DESCRIPTION:
In this study, it was aimed to investigate the effect of Ultrasound guided superficial cervical plexus block versus greater auricular nerve block for on postoperative tympanomastoid surgery analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class and underwent Tympanomastoid surgery.

Exclusion Criteria:

* Previous history of opioid use preoperatively,
* Allergy to local anesthetics,
* The presence of any systemic infection,
* Uncontrolled arterial hypertension,
* Uncontrolled diabetes mellitus.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | Postoperative 24 hours
  Visual Analog Pain Scale was used for pain

SECONDARY OUTCOMES:
tramadol consumption | Postoperative 24 hour
  tramadol consumption
side effect profile | Postoperative 24 hour
  side effect profile (including nausea and vomiting, hypotension,requirement and the Ramsay Sedation Scale (RSS) scores)
additional analgesic use | Postoperative 24 hour
  additional analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, M.D, Principal Investigator — University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospita